CLINICAL TRIAL: NCT00319605
Title: Cross Sectional Study to Evaluate the Acceptability of Oral Solution of Levetiracetam (Keppra®) (SOLUCION Study)
Brief Title: Cross Sectional Study to Evaluate the Acceptability of Oral Solution of Levetiracetam
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: N01242
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Epilepsy
Keywords: Cross sectional study; acceptability; levetiracetam; oral solution; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
Phase IV, observational, post-authorization, cross sectional, open-label, multicenter study to evaluate the acceptability of oral solution of levetiracetam in patients with partial epilepsy as assessed by a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients 16 years old or older diagnosed with partial epilepsy with or without generalization receiving levetiracetam oral solution for at least 28 days before the study

Exclusion Criteria:

* Patients with disturbances of the sense of taste and smell that can interfere with the assessment of the parameters of the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study populaton is defined. See Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Marin Muñoz, MD, Study Director — UCB Pharma
Locations (54):
- Spain (54):
  - A Coruña
  - Alcalá de Henares
  - Alcázar de San Juan
  - Alcorcón
  - Alicante
  - Alzira Valencia
  - Ávila
  - Badajoz
  - Barcelona
  - Benidorm
  - Cadz
  - Castellon
  - Cáceres
  - Cuenca
  - Elda
  - Eliana
  - Girona
  - Granada
  - Guadalajara
  - Hospitalet Del Llobregat
  - La Roca
  - Langreo
  - Las Palmas
  - Las Palmas de Gran Canaria
  - León
  - Lleida
  - Lorca Murcia
  - Lugo
  - Madrid
  - Manzanares
  - Manzanares Ciudad Real
  - Mataró
  - Málaga
  - Merida Badajoz
  - Móstoles
  - Murcia
  - Oviedo
  - Palencia
  - Palmar
  - Pamplona
  - Pontevedra
  - Puerto del Rosario
  - Sabadell
  - Salamanca
  - San Fernando
  - Santa Cruz de Tenerife
  - Seville
  - Terrassa
  - Teruel
  - Toledo
  - Valencia
  - Vigo Pontevedra
  - Zamora
  - Zaragoza